CLINICAL TRIAL: NCT06889090
Title: Comparing Effect of Opioid-sparing Versus Conventional Anesthesia on Quality of Recovery After Emergency Laparotomy: a Randomized Controlled Trial
Brief Title: Comparing Effect of Opioid-sparing Versus Conventional Anesthesia on Quality of Recovery After Emergency Laparotomy
Acronym: O-S Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Madkour, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ty7890567
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia Recovery Period
MeSH Terms: interventions — Syringes; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- opioid sparing (Active Comparator): two syringes of lidocaine 10 mg/mL will be prepared. A 10-mL syringe (induction syringe) will be given during the induction of anesthesia and A 50 mL syringe (infusion syringe) will be used as continuous infusion.
  Interventions: Drug: : two syringes of lidocaine 10 mg/mL will be prepared. A 10-mL syringe (induction syringe) will be given during the induction of anesthesia and A 50 mL syringe (infusion syringe) will be used as conti
- conventional (Placebo Comparator): A 10-mL syringe of 10 mcg/mL fentanyl (induction syringe) and a 50-mL syringe of saline (infusion syringe) will be prepared as placebo.
  Interventions: Drug: A 10-mL syringe of 10 mcg/mL fentanyl (induction syringe) and a 50-mL syringe of saline (infusion syringe) will be prepared as placebo.

INTERVENTIONS:
Drug: : two syringes of lidocaine 10 mg/mL will be prepared. A 10-mL syringe (induction syringe) will be given during the induction of anesthesia and A 50 mL syringe (infusion syringe) will be used as conti — : two syringes of lidocaine 10 mg/mL will be prepared. A 10-mL syringe (induction syringe) will be given during the induction of anesthesia and A 50 mL syringe (infusion syringe) will be used as continuous infusion.
  Arms: opioid sparing
Drug: A 10-mL syringe of 10 mcg/mL fentanyl (induction syringe) and a 50-mL syringe of saline (infusion syringe) will be prepared as placebo. — A 10-mL syringe of 10 mcg/mL fentanyl (induction syringe) and a 50-mL syringe of saline (infusion syringe) will be prepared as placebo.
  Arms: conventional

SUMMARY:
Aim of the Work The investigators aim to compare lidocaine-based anesthesia versus conventional anesthesia in the presence of multimodal analgesia protocol in terms of early quality of recovery and analgesic efficacy.

Objectives To compare quality of recovery using the Quality of recovery-15 (QoR-15) score between lidocaine-based anesthesia in relation to conventional anesthesia in patients undergoing emergency laparotomy.

Hypothesis the investigators hypothesize that lidocaine-based regimen would be effective in reducing opioid use and provide superior quality of recovery compared to conventional opioid-routine anesthesia in emergency laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-65 years)
* ASA I-III undergoing emergency laparotomy with midline incision.

Exclusion Criteria:

* Severe cardiac morbidities (impaired contractility with ejection fraction < 45%, heart block, arrhythmias, tight valvular lesions) and patients on beta-blockers
* Patients on vasopressor infusion, patients with high shock index (heart rate / systolic blood pressure >1)
* Body mass index <18 or > 35 Kg/m2,

  * Pregnant or lactating women,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
- Quality of recovery using the QoR-15 score 24 h after surgery. | 24 hours
  - Quality of recovery using the QoR-15 score 24 h after surgery. An 11-point numerical rating scale (for positive items, 0 = "none of the time" to 10 = "all of the time"; for negative items the scoring was reversed; maximum score 150).

IPD SHARING:
Plan to Share IPD: No